CLINICAL TRIAL: NCT01233765
Title: Analysis of Neutrophil Response in Chronic Periodontitis (Including the Project Entitled 'Pro-Inflammatory Cytokine Production by Neutrophils in Periodontitis Patients')
Brief Title: Analysis of Neutrophil Response in Chronic Periodontitis
Status: Completed | Type: Observational
Sponsor: Birmingham Community Healthcare NHS (Other Government)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Professor I Chapple, Professor (PI), Birmingham Community Healthcare NHS
Other Study IDs: RG_10-077
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Chronic Periodontitis
Keywords: Periodontitis; Neutrophil; Inflammation
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control volunteers with periodontal health: Control volunteers with periodontal health
- Patient volunteers with chronic periodontitis: Patient volunteers with chronic periodontitis

SUMMARY:
Recent scientific evidence suggests that the main defence cell of the body (neutrophil) behaves in a different manner in patients with gum disease; namely how they interact with bacteria and their role in defence systems of the body. This study proposes to examine these responses in periodontitis patients and healthy controls.

The proposed study will include patients undergoing periodontal (gum) treatment who will be matched to periodontally healthy controls. Blood, gingival crevicular (gum) fluid and clinical measures will be collected both pre- and post-therapy to measure differences in cell behaviour both before, and following routine therapy.

Blood samples will be used to isolate peripheral blood neutrophils prior to analysis of their responses to different bacterial stimuli including oxygen radical, cytokine and extracellular trap release. Gingival Crevicular Fluid samples will be used to measure different biochemical markers that result from the production of Neutrophil Extracellular Traps (NETs). Routine clinical measures will be taken both pre- and post-therapy as a measure of treatment response.

Patient volunteers undergoing treatment will be asked to donate a total of four small samples of tissue from the gums whilst they are already anaesthetised for routine treatment. These will be approximately the size of a needle head (2mm2mm) and used to examine NET formation within the tissues and related processes. This will provide novel in-vivo data regarding this recently discovered method of neutrophil defence in innate immunity.

This proposal represents a novel study aimed at improving our current understanding of why inflammatory periodontitis develops in some patients but not others, as well as providing pointers to causal/noncausal relationships between periodontitis and important systemic conditions such as diabetes and rheumatoid arthritis.

Ultimately, novel treatment approaches and primary prevention (for periodontitis) or secondary prevention (for systemic disease) strategies may emerge.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 or over
* Have a minimum of 20 teeth
* Have chronic periodontitis or otherwise healthy volunteers (controls)
* Be capable of giving informed consent themselves and are able and willing to participate in the study

Exclusion Criteria:

* Patients with aggressive disease
* Mouthwash use
* Special dietary needs (e.g. coeliac)
* Patients with physical or mental disability
* Pregnant women or those breastfeeding
* Patients whose medical history may place them at risk of complications from periodontal therapy (e.g. warfarinised volunteers)
* Patients taking long term anti-microbial or anti-inflammatory drugs
* Patients unable or unwilling to provide informed consent
* Taking dietary supplements (e.g. multivitamins, antioxidants, fish oils)
* Shows unwillingness, inability or lack of motivation to carry out the study procedures, or cannot conform to the protocol
* A course of antibiotic or anti-inflammatory therapy currently or in the previous 3 months
* Current orthodontic treatment (e.g. wearing braces or orthodontic devices)
* Currently participating in another dental trial
* Diabetics
* Smokers or have smoked up to within 5 years
* Those patients who disclose previous or current recreational drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will comprise 20 competent adult volunteers (>18 years old) recruited from patients attending for clinical examination following referral for a specialist opinion for periodontal disease, and will be recruited on the basis of clinical need. In addition, 20 periodontally-healthy controls will be recruited from staff or students of the School of Dentistry and Biomaterials and Birmingham Dental Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Principal Research Question | Three months for each matched patient and control
  Do leukocyte (neutrophil) responses differ between patients diagnosed with periodontitis compared to matched healthy controls, and what is the effect of standard periodontal treatment and stabilisation on this response?

SECONDARY OUTCOMES:
Secondary Research Question | Three months for each matched patient and control
  Can markers of the white blood defence cells (neutrophils) be observed and measured in-vivo within the local tissues and if so do they differ between inflamed and non-inflamed sites?

CONTACTS AND LOCATIONS:
Locations (1):
- University of Birmingham School of Dentistry, Birmingham, West Midlands, United Kingdom